CLINICAL TRIAL: NCT03067376
Title: An Open-label, Single-dose Study Designed to Assess the Mass Balance Recovery, Metabolite Profile and Identification of Metabolite Structures for [14C]-CORT125134 in Healthy Subjects
Brief Title: A Study Designed to See How [14C]-CORT125134 is Taken up, Broken Down and Removed From the Body
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CORT125134-121; 2016-000668-41 (EudraCT Number)
Record Dates: First submitted 2016-12-06; First posted 2017-03-01 (Actual); Last update posted 2019-08-09 (Actual); Status verified 2019-08

CONDITIONS: Healthy
Keywords: Absorption, distribution, metabolism, and excretion (ADME); Metabolism; Metabolite Profiling; Excretion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [14C]-CORT125134 (Experimental): Two capsules each containing 125 milligrams (mg) [14C]-CORT125134 administered to each participant on 1 occasion
  Interventions: Drug: [14C]-CORT125134

INTERVENTIONS:
Drug: [14C]-CORT125134

SUMMARY:
The study was designed to evaluate how CORT125134 is taken up, broken down and removed from the body when given as an oral capsule to healthy subjects.

DETAILED DESCRIPTION:
The study was conducted to determine the recovery of [14C]-CORT125134 after the administration of a single oral dose of [14C]-CORT125134, to determine the routes and rate of elimination of [14C]-CORT125134 and associated radioactivity from the body, and to measure concentrations of radioactivity in the blood. Additional objectives of the study were to determine the chemical structure of each significant metabolite in plasma, urine and feces. Safety and tolerability were assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or healthy females of non-childbearing potential (surgically sterilized or postmenopausal [defined as a woman of with at least a 12 month history of amenorrhea with a follicle-stimulating hormone (FSH) >40 international units per liter (IU/L) in the absence of a reversible medical iatrogenic cause])
* Age 30 to 65 years of age
* A history of regular bowel movements (averaging ≥1 and ≤3 stools per day)
* Must be willing and able to communicate and participate in the whole study
* Must provide written informed consent
* Male participants must agree to use an adequate method of contraception
* Participants are willing to abide by the study restrictions

Exclusion Criteria:

* Participation in a clinical research study within the previous 3 months
* Participants who have previously been enrolled in this study or participants who have previously been treated with CORT125134
* History of any drug or alcohol abuse in the past 2 years
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 milliliter (mL) of 40% spirit or a 125 mL glass of wine)
* Current smokers and those who have smoked within the last 12 months; this includes cigarettes, e-cigarettes and nicotine replacement products. A breath carbon monoxide reading of greater than 10 parts per million (ppm)
* Females of childbearing potential (female participants must have a negative urine pregnancy test)
* Male Participants with pregnant partners
* Radiation exposure exceeding 5 millisievert (mSv) in the last 12 months or 10 mSv in the last 5 years. The measurement includes exposure from the present study, and diagnostic x rays and other medical exposures, but excludes background radiation. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 1999.
* Positive drugs of abuse test result
* Participants who are taking, or have taken, any prescribed or over-the-counter drug (other than 4 grams per day paracetamol) or herbal remedies in the 14 days before study drug administration. Hormone replacement therapy is not permitted

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2016-08; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Amount of radioactivity eliminated in urine | Day 1 pre-dose to Day 8 post-dose
Amount of radioactivity eliminated in feces | Day 1 pre-dose to Day 8 post-dose
Amount of radioactivity eliminated in urine and feces | Day 1 pre-dose to Day 8 post-dose
Cumulative amount of radioactivity eliminated in urine | Day 1 pre-dose to Day 8 post-dose
Cumulative amount of radioactivity eliminated in feces | Day 1 pre-dose to Day 8 post-dose
Cumulative amount of radioactivity eliminated in urine and feces | Day 1 pre-dose to Day 8 post-dose
Pharmacokinetics (PK) of total radioactivity: lag time (tlag) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: peak plasma concentration (Cmax) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: time to reach maximum observed concentration (tmax) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: area under the plasma concentration-time curve from time zero to time of last measurable concentration (AUClast) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: area under the plasma concentration-time curve from time zero to infinity (AUCinf) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: area under the plasma concentration-time curve extrapolated from time t to infinity as a percentage of total AUC (%AUCextrap) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: first-order elimination rate constant associated with the terminal portion of the curve, determined as the negative slope of the terminal log-linear phase of the drug concentration-time curve (lambda-z) | Day 1 pre-dose to Day 8 post-dose
PK of total radioactivity: elimination half-life (t1/2) | Day 1 pre-dose to Day 8 post-dose
Metabolic profiling and structural identification in plasma, urine and feces | Day 1 pre-dose to Day 8 post-dose

SECONDARY OUTCOMES:
Hematology | Screening, Day 1 pre-dose, Day 8
Clinical chemistry | Screening, Day 1 pre-dose, Day 8
Urinalysis | Screening, Day 1 pre-dose, Day 8
Blood pressure | Screening, Day 1 pre-dose and 2 hours post-dose, Day 8
Heart rate | Screening, Day 1 pre-dose and 2 hours post-dose, Day 8
Electrocardiogram | Screening, Day 1 pre-dose and 2 hours post-dose, Day 8
Percentage of subjects with adverse events | Screening to Day 28
Physical examination | Screening and Day 8
Tlag of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Cmax of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Tmax of CORT125134 | Day 1 pre-dose to Day 8 post-dose
AUClast of CORT125134 | Day 1 pre-dose to Day 8 post-dose
%AUCextrap of CORT125134 | Day 1 pre-dose to Day 8 post-dose
AUCinf of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Lambda-z of CORT125134 | Day 1 pre-dose to Day 8 post-dose
T1/2 of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Mean Residence Time (MRT) of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Apparent oral clearance (CL/F) of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Apparent volume of distribution (Vz/F) of CORT125134 | Day 1 pre-dose to Day 8 post-dose
Number of metabolites >10% of circulating radioactivity in plasma | Day 1 pre-dose to Day 8 post-dose
Number of metabolites >10% of the dose in urine | Day 1 pre-dose to Day 8 post-dose
Number of metabolites >10% of the dose in feces | Day 1 pre-dose to Day 8 post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, MBChB, Principal Investigator — Quotient Clinical
Locations (1):
- Quotient Clinical, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No